CLINICAL TRIAL: NCT06258187
Title: Randomized Control Trial of Colorimetric CO2 Detectors for Ventilation Assessment in the Delivery Room
Brief Title: Pedi-Cap CO2 Detector for Face-mask Ventilation in the Delivery Room
Acronym: CO2-Vent
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Riti Chokshi, MD, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: STU-2023-0969
Record Dates: First submitted 2024-01-15; First posted 2024-02-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Neonatal Resuscitation; Neonatal Disease
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Intervention Model Description: The quasi-randomization scheme will be determined by a non-investigator for each month. This will be revealed at the beginning of each month on whether to use Pedi-Cap or not during delivery room resuscitation using sealed, opaque envelopes.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Pedi-Cap (Experimental): A Pedi-Cap will be connected to the T-piece resuscitator in between the T-piece and face mask. With effective gas exchange, carbon dioxide (CO2) is detected by the Pedi-cap and will demonstrate gold color change with each exhalation. If there is no CO2 gas exchanged, the Pedi-Cap color will remain purple. The color change will be used as one of the tools for the resuscitation team to determine if the infant has effective non-invasive positive pressure ventilation (PPV) during delivery room resuscitation. Other ways, in addition to the Pedi-Cap, to determine effective PPV include a rise in heart rate, improved infant color, chest rise, and improvement in oxygen saturation.
  Interventions: Device: Pedi-Cap
- No Pedi-Cap (No Intervention): There will be no Pedi-Cap attached to the t-piece resuscitator. Effective non-invasive positive pressure ventilation (PPV) during delivery room resuscitation will be assessed by a rise in heart rate, improved infant color, chest rise, and improvement in oxygen saturation.

INTERVENTIONS:
Device: Pedi-Cap — The neonatal resuscitation team will include or omit the use of Pedi-Cap during non-invasive positive pressure ventilation (PPV) for infants ≥30 weeks in the delivery room based on the randomized study arm each month.
  Other Names: Colorimetric carbon dioxide (CO2) detector
  Arms: Pedi-Cap

SUMMARY:
The goal of this study is to determine if using a Pedi-Cap (a type of colorimetric carbon dioxide detector) during face mask ventilation (PPV) for newborn infants in the delivery room will lower the time of PPV needed. A group of nurses, doctors, and respiratory therapists, called the neonatal resuscitation team, will either use or not use the Pedi-Cap during face mask PPV for infants born at ≥30 weeks' gestation.

A randomization generator will assign each month to either use the Pedi-Cap or not use the Pedi-Cap. The researchers will collect information from the medical chart to find the infant and mother's information, medical interventions done in the delivery room, and lab values. In addition, resuscitation team members will fill out a survey of their experiences of using or not using the Pedi-Cap during delivery room facemask PPV.

DETAILED DESCRIPTION:
This is an open, prospective, quasi-randomized, single center trial that will address the primary research question: Does use of a colorimetric carbon dioxide (CO2) detector (Pedi-Cap) decrease the duration of non-invasive positive pressure ventilation (PPV) in the delivery room? The neonatal resuscitation team, comprised of nurses, doctors, and respiratory therapists will include or omit the Pedi-Cap during noninvasive PPV for infants born at ≥30 weeks' gestation in the delivery room. The quasi-randomization scheme will be determined by a opening an opaque envelope each month. This will be revealed at the beginning of each month on whether to use the Pedi-Cap or not. Other outcomes variables that will be assessed include initial heart rate (HR), time to HR > 100 bpm, duration of bradycardia, time to start of ventilation corrective maneuvers (if needed), maximum peak inspiratory pressure used, maximum peek inspiratory pressure used, maximum fractionated inspired oxygen, time to gold color change on Pedi-Cap, need for intubation, need for delayed PPV, need for chest compressions/epinephrine, need for neonatal intensive care unit admission if infant ≥35 gestational age, occurrence of pneumothorax, length of mechanical ventilation in days, doses of surfactant given, and survival to discharge. Infant and maternal characteristics will be obtained from the electronic medical record. Association of outcomes with each study arm will be stratified by infant and maternal characteristics.

In addition, a survey will be administered to the resuscitation team members at the completion of the study to assess their experience with each study arm.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at ≥30 weeks' gestation
* Presence of the resuscitation team prior to delivery
* Need for non-invasive positive pressure ventilation (PPV).

Exclusion Criteria:

* Infants born at <30 weeks' gestation
* No non-invasive PPV needed in the delivery room
* Infants with conditions requiring immediate intubation such as congenital diaphragmatic hernia
* Resuscitation team not present prior to delivery/need for PPV
* Infants who have a prenatal plan of comfort care only

Min Age: 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 632 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Duration of positive pressure ventilation (PPV) | From birth to end of delivery room resuscitation or admission to the Neonatal Intensive Care Unit (NICU) (approximately 1 hour of life)
  The time that an infant needs non-invasive PPV during delivery room resuscitation.

SECONDARY OUTCOMES:
Duration of bradycardia | From birth to end of delivery room resuscitation or admission to the NICU (approximately 1 hour of life)
  The time that an infant has a heart rate of less than 100 beat per minute during delivery room resuscitation.
Time to heart rate great than 100 beats per minute | From birth to end of delivery room resuscitation or admission to the NICU (approximately 1 hour of life)
  The ultimate goal of a successful delivery room resuscitation is to sustain the infant's heart rate above 100 beats per minute.
time to start of ventilatory corrective maneuvers | From birth to end of delivery room resuscitation or admission to the NICU (approximately 1 hour of life)
  As per the neonatal resuscitation program algorithm 8th edition, if the infant's heart rate does not improve with non-invasive ventilation, corrective steps must be taken to optimize non-invasive ventilation such as suctioning, repositioning, adjusting the mask, opening the mouth/nose, and increasing the peak inspiratory pressure.
Maximum peak inspiratory pressure used | From birth to end of delivery room resuscitation or admission to the NICU (approximately 1 hour of life)
  As per the neonatal resuscitation program algorithm 8th edition, if the infant's heart rate does not improve with non-invasive ventilation, corrective steps must be taken to optimize non-invasive ventilation such as increasing peak inspiratory pressure.
Time to gold color change on Pedi-Cap | From birth to end of delivery room resuscitation or admission to the NICU (approximately 1 hour of life)
  Gold color change on the Pedi-Cap indicates carbon dioxide (CO2) exchange occurring and correlates with increased tidal volumes and increased heart rate.
Need for intubation in the delivery room | From birth to end of delivery room resuscitation or admission to the NICU (approximately 1 hour of life)
  Need for intubation as per the neonatal resuscitation program algorithm 8th edition if the infant's heart rate does not improve with non-invasive ventilation.
need for delayed positive pressure ventilation | From birth to end of delivery room resuscitation or admission to the NICU (approximately 1 hour of life)
  Need for a subsequent positive pressure ventilation after an initial cessation
Need for chest compressions or epinephrine | From birth to end of delivery room resuscitation or admission to the NICU (approximately 1 hour of life)
  Need for chest compression and epinephrine as per the neonatal resuscitation program algorithm 8th edition if the infant's heart rate does not improve with invasive ventilation.
Need for neonatal intensive care unit admission if infant ≥35 gestational age | From birth to end of delivery room resuscitation or admission to the NICU (approximately 1 hour of life)
  Generally, infants born ≥35 gestational age are not admitted to the neonatal intensive care unit unless there are delivery room complications or neonatal disease.
Occurrence of pneumothorax | From birth to 3 days of life
  The risk of positive pressure ventilation can be a pneumothorax.
Duration of mechanical ventilation | From birth to date of discharge or death, whichever comes first, assessed up to 50 weeks
  The number of days and infant requires mechanical ventilation
Need for surfactant | From birth to date of discharge or death, whichever comes first, assessed up to 50 weeks
  The need for surfactant administration
Maximum positive end expiratory pressure used | From birth to end of delivery room resuscitation or admission to the NICU (approximately 1 hour of life)
  As per the neonatal resuscitation program algorithm 8th edition, if the infant does not have good oxygen saturation, interventions must be done to meet goal saturations for each minute of life.
Maximum fractionated inspired oxygen used | From birth to end of delivery room resuscitation or admission to the NICU (approximately 1 hour of life)
  As per the neonatal resuscitation program algorithm 8th edition, if the infant does not have good oxygen saturation, interventions must be done to meet goal saturations for each minute of life.
Survival to discharge | birth to discharge from NICU (up to 12 months of age)
  Determination if the infant is discharged home

OTHER OUTCOMES:
Initial heart rate at birth | From birth to initial assessment by resuscitation team members (approximately by 2 minutes of life)
  The initial heart rate in beats per minute at the first recording after birth

CONTACTS AND LOCATIONS:
Overall Officials: Riti Chokshi, Principal Investigator — University of Texas
Locations (1):
- Parkland Health, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wyckoff MH, Wyllie J, Aziz K, de Almeida MF, Fabres J, Fawke J, Guinsburg R, Hosono S, Isayama T, Kapadia VS, Kim HS, Liley HG, McKinlay CJD, Mildenhall L, Perlman JM, Rabi Y, Roehr CC, Schmolzer GM, Szyld E, Trevisanuto D, Velaphi S, Weiner GM; Neonatal Life Support Collaborators. Neonatal Life Support: 2020 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2020 Oct 20;142(16_suppl_1):S185-S221. doi: 10.1161/CIR.0000000000000895. Epub 2020 Oct 21. PMID 33084392
- [Background] Perlman JM, Wyllie J, Kattwinkel J, Atkins DL, Chameides L, Goldsmith JP, Guinsburg R, Hazinski MF, Morley C, Richmond S, Simon WM, Singhal N, Szyld E, Tamura M, Velaphi S; Neonatal Resuscitation Chapter Collaborators. Neonatal resuscitation: 2010 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science with Treatment Recommendations. Pediatrics. 2010 Nov;126(5):e1319-44. doi: 10.1542/peds.2010-2972B. Epub 2010 Oct 18. No abstract available. PMID 20956431
- [Background] Weiner MDFGM. NRP Textbook of Neonatal Resuscitation. 8th. ed. Itasca: American Academy of Pediatrics; 2021.
- [Background] ILCOR Summary Statement: 2023 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science with Treatment Recommendation 2023 [Available from: https://ilcor.org/publications/preprint